CLINICAL TRIAL: NCT02829632
Title: 12 Weeks Weight Loss Study Using Feedback Messages Delivered Via Smartphone
Brief Title: Feasibility Study of Receiving Feedback Messages Based on Self-monitored Dietary Intake
Acronym: SMARTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Lora Burke, Professor of Nursing and Epidemiology, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PRO14110537
Record Dates: First submitted 2015-07-02; First posted 2016-07-12 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Overweight; Obesity
Keywords: mobile technology; feedback message; self-monitoring
MeSH Terms: conditions — Overweight; Obesity | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental: Group Sessions (Experimental): Participants will be asked to attend 3 group meetings over a 12 week period. Groups will meet for approximately 1 hour on weeks 2, 4 and 8. At each of the group meetings, the participant will be weighed and a group leader will present information on topics related to eating and exercise.
  Interventions: Behavioral: Group Sessions; Behavioral: Feedback; Behavioral: Self-monitoring
- Active Comparator: Self-Monitoring (Experimental): Active Comparator: Self-monitoring Participants will record diet, activity and weight as described above in the participant's smartphone app to assist the participant in losing weight.
  Interventions: Behavioral: Self-monitoring
- Experimental: Feedback (Experimental): Participants will be sent via the participant's smartphone between
  1 and 4 feedback messages a day about whether the participant has been self monitoring, or the amount of calories, fat or sugar the participant has consumed.
  Interventions: Behavioral: Feedback; Behavioral: Self-monitoring

INTERVENTIONS:
Behavioral: Group Sessions — Participants will receive a 3-session behavioral lifestyle program for a healthful lifestyle and weight loss.
  Arms: Experimental: Group Sessions
Behavioral: Feedback — Participants will receive up to 4 daily feedback messages based on progress in attaining target behavior. The feedback messages will be delivered on a variable ratio schedule and tailored to data in subjects' dietary recordings.
  Arms: Experimental: Feedback; Experimental: Group Sessions
Behavioral: Self-monitoring — Participants will receive an one-time how to self-monitor using the smartphone session.

SUMMARY:
Brief Summary: This randomized clinical pilot will test the feasibility of having individuals self-monitor for 12 weeks and based on what the participants record be given feedback messages. The investigator will use this information to refine the questions and data collection procedures for the larger study.

Participants will be randomized into 3 groups

* self-monitoring only
* self-monitoring w/ feedback messages
* self-monitoring w/feedback messages and group sessions Feedback messages will be delivered up to 4 times per day using a different schedule. The group sessions will be held in the 2nd, 4th and 8th week of the 12-week study.

All participants will be asked to complete questionnaires and 2 assessment visits at baseline and 12 weeks.

DETAILED DESCRIPTION:
Research Strategy. The investigator will randomize 45 overweight/obese adults to one of 3 groups: (1) Control (Con) - no FB, no Behavioral Lifestyle Program (BLP), (2) FB Only, no BLP, and (3) FB+BLP. All subjects will use a smartphone to self-monitor diet and PA. The subjects will download a feedback system onto the Android operating system smartphone that was developed for this study called the SMARTER. The algorithm was developed by Dr. Lora Burke of the University of Pittsburgh. All groups will attend a one-time how to self-monitor using the smartphone session and receive education materials at baseline. The FB Only and FB+BLP groups will receive up to 4 daily FB messages, based on progress in attaining target behavior. The FB will be delivered on a variable ratio schedule and tailored to data in subjects' recordings. FB+BLP participants will receive a face-to-face BLP intervention that will include 3 group sessions over 12 weeks. Also to not confound the effect of the daily FB, the interventionists will not provide feedback to the weekly diaries. Sample. The investigator will recruit from the community 45 adults, over the age of 18. All participants need to be randomized prior to the beginning of the 3 BLP sessions since the sessions are conducted as a closed group. The randomization scheme will be implemented via a computerized program (Visual Basic 6.0) using minimization method. The randomization will be overseen by a statistician (Co-I: S Sereika). Each of the 3 conditions will be assigned a total of 15 subjects with randomization stratified by gender and ethnicity/race. Intervention. Those in the Con and FB Only groups will receive a 1-hr session on provided calorie prescription for weight loss and self-monitoring and associated education materials. Only those in FB+BLP will receive a 3-session BLP for a healthful lifestyle and weight loss. The groups will meet in the School of Nursing and will be led by a trained interventionist. Protocol for Self-monitoring: All participants will be subscribed to LoseIt!, an online self-monitoring service that can be accessed via the smartphone and computer. This will be used in place of the traditional paper diary. This software permits self-monitoring of diet, PA, and weight; it also provides feedback on up to 9 macronutrients based on a database of 60,000 foods. Because of the investigator's ongoing working relationship with the developers of LoseIt! program, the investigator will have access to LoseIt! Connect, a custom portal created by LoseIt! for centralized user management. This permits the investigators to view participants' entries and set custom controls on participants use, (e.g., disabling particpants' ability to share data with outsiders). All participants will be encouraged to self-monitor diet and self-report weight. Participants who do not have scales will be given one for the duration of the study and be ask to return it at the completion of the study. Participants see the nutrient value of each food and the calculated subtotals. The interventionists will have access to the diaries so participants can contact a participant if there is any concern about the reported eating behaviors. This is the same procedure used for the past 4 years in the EMPOWER Study (IRB - PRO10100504). At the training session, participants will be advised on how to change the privacy settings on Lose It!. General Information about Feedback Algorithm. The FB algorithm programmed in the FB app will use real-time synced self- monitoring data to send messages that are responsive to the participants' entries. The server will deliver a message that will be displayed on the screen of the smartphones so the person does not need to make extra clicks to view it. The FB messages will address one target behavior at a time, e.g., self-monitoring or calorie intake. At the baseline education session for the FB Only group or the first BLP session for FB+BLP, the individual will make a diary entry; the system will send a FB message shortly thereafter to provide immediate reinforcement for self-monitoring. Then the FB will be delivered on the incremental 1-4 x/d schedule, contingent on progress in self-monitoring and in attaining the person's daily calorie goal. Rules will be applied to the delivery of messages to FB Only and FB+BLP, e.g., messages will be delivered between the hours set by the participants on particpants phone, e.g., 8 AM and 9:30 PM, and content will be guided by the parameters built into the algorithm. In the implementation of the proposed FB intervention, the investigators will exercise caution and sensitivity regarding participants' reception of the messages. In the SMART Trial, the messages were motivating and reinforcing, not noting deficiencies in behavior or progress not made; however, the messages will provide guidance for corrective action when the person is not following the behavior that would be consistent with the pre-established goals. Space does not permit extensive message samples but examples might be as follows. Excellent job on increasing fruits in your diet. OR Super job staying within the fat limits. Go easy on high fat foods tonight; consider having a big salad with nonfat dressing. Protocol for the Behavioral Lifestyle Program (BLP) intervention: Group Sessions: Participants will receive nutritional and behavioral counseling; practical hands-on experiences to develop skills to implement a healthy lifestyle (e.g., practice mindful eating, portion size, modify foods or meals to reduce fat content) in three 1 hour group sessions. The groups will meet evenings and will be led by the multidisciplinary team (behavioral scientists, nutritionists that has been trained by the PI and Co-I (Burke and Ewing). The group sessions will be held in the 2nd, 4th and 8th week of the 12-week study. Behavior Goals: Calorie: The calorie goal will be calculated from the individual's baseline body weight (1200 - 1800 kcal for <250 lbs or 1800 to 2000 kcal for >250 lbs). Calorie goals can be adjusted if necessary for participants struggling to meet the goa;s or for maintenance. Fat: Fat gram goals will 40 - 60 grams per day depending on calorie goal. Screening Measures - administered only at baseline. Sociodemographic Form will be used to collect data on individual characteristics, e.g., ethnicity, marital status. Rapid Eating Assessment for Patients (REAP) will be used to assess current diet to inform the goals for lifestyle improvement. It has 31 items that ask about weight, PA and sedentary habits, variety in diet, excess food intake. Participants Online Screening Questionnaire will be used to assess Qualtric systems as a screening tool. It will be given with the other screening questionnaires at their Baseline Assessment. Outcome or Dependent Measures. Unless otherwise noted, all measures will be conducted at 0 and 12 weeks. Trained staff will perform these in the Clinical Research Suite in the School of Nursing. Participants will be compensated for completing the 12-week assessment. BMI- Weight - measured with the Tanita Scale and Body Fat Analyzer with subjects in light clothing standing bare foot on the scale's footpads. Height (centimeters) measured with stadiometer for BMI (kg/m2) calculation. Cardiometabolic risk factors Blood pressure (BP). BP assessment will follow the standard AHA guidelines and measured using an Omron BP Monitor with ComFit cuff with the subject in a sitting position after at least a 5-min rest. Whole body composition. To describe % fat mass, we will measure body composition (fat mass, % fat, fat-free mass) by bioelectrical impedance analysis on the Tanita Scale and Body Fat Analyzer.120 Waist circumference will be measured twice with a Gullick II measuring tape. If the two values are within 2 cm of each other, a mean is calculated; if not, measurements are taken again until they are within 2 cm. Psychosocial surveys.

Weight Efficacy Lifestyle (WEL) is a 20-item scale used to assess level of confidence to resist eating in varied situations or emotional states. It has established psychometric properties 135 and takes 5 min to complete. This scale has added explanatory value in weight loss behavior in our previous studies. The Newest Vital Sign, a brief test of literacy applied to reading a food label. At the completion of study, the groups that were not randomized into the group sessions will receive the session material via email.

The group that did not receive feedback messages will be given the option of receiving messages for 12 weeks. If the participant chooses to have the feedback messages, it will be loaded on the participant's phones at the 12 weeks assessment.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* BMI between 27-43
* have an Android smartphone,
* has not used app for self-monitoring at least 4 days/week for the past 3 months
* can attend group meetings.

Exclusion Criteria:

* persons who plan to become pregnant
* have diabetes or a medical condition in which weight loss in contraindicated
* unable to walk for exercise
* on a weight loss drug
* had bariatric surgery
* plans to relocate within 3 months of recruitment
* currently in a weight loss program. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in weight | 12 weeks
  Changes in weight: measured as Percent change in weight from baseline to 12 weeks

SECONDARY OUTCOMES:
Adherence to treatment protocol | 12 weeks
  Number of days participants self-monitor
Adherence to self-weighing protocol | 12 weeks
  Number of days participants self-weigh

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
there is no plan to share the data. The data are being used for a grant application.

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882